CLINICAL TRIAL: NCT03884179
Title: Diagnosis of Pancreatic Cystic Lesions With EUS-FNA and Cross-sectional Imaging - A Report of Accuracy
Brief Title: Diagnosis of PCL With EUS-FNA and Cross-sectional Imaging - A Report of Accuracy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Riadh Sadik, Ass Prof, Sahlgrenska University Hospital
Other Study IDs: SahlgrenskaUHGEA2017
Record Dates: First submitted 2018-04-24; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cyst; Pancreatic Neuroendocrine Carcinoma; Pancreatic Pseudocyst; Pancreatic Serous Cystadenoma; Pancreatic Mucinous Cystadenoma; Pancreatic Cystadenocarcinoma; Pancreatic Intraductal Papillary-Mucinous Neoplasm; Solid Pseudopapillary Tumor of the Pancreas
Keywords: Endoscopic ultrasound; Radiology; Accuracy; Pancreatic Cyst; Pancreatic Cystadenocarcinoma; Pancreatic Mucinous Cystadenoma; Pancreatic Intraductal Papillary-Mucinous Neoplasm; Pancreatic Serous Cystadenoma; Pancreatic Pseudocyst; Pancreatic Neuroendocrine Tumor; Solid Pseudopapillary Tumor of the Pancreas
MeSH Terms: conditions — Pancreatic Cyst; Somatostatinoma; Pancreatic Pseudocyst; Pancreatic Intraductal Neoplasms; Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cystic lesions (PCLs) comprise of a heterogeneous group of entities that are benign, premalignant or malignant. With increased use of modern imaging techniques in recent years, incidentally discovered PCL have become much more common. However, imaging modalities for characterising PCL is a known clinical uncertainty since imaging is capable of detecting these lesions but may often not be able to distinguish malignant from benign lesions. Incorrect assessment of PCL can lead to fatal consequences because a malignant lesion may not be treated and a benign may be unnecessarily resected. The aim of this study was to assess the performance of endoscopic ultrasound with fine-needle aspiration (EUS-FNA) in the diagnosis of pancreatic cystic lesions compared to cross-sectional imaging modalities (CT/MRI). Our hypothesis is that EUS-FNA has a higher accuracy for diagnosing PCLs compared with cross-sectional imaging.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected PCLs according to radiology undergoing evaluation with EUS-FNA at a tertiarry endoscopy center from February 2007 until March 2017, who underwent pancreas resection

Oral and written consent of patients examined

Exclusion Criteria:

None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected PCLs according to radiology undergoing evaluation with EUS-FNA at a tertiarry endoscopy center from February 2007 until March 2017. The catchemnt area of this cente has a population of about two million.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2007-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of EUS-FNA vs Radiology | 10 years
  To compare the accuracy of EUS-FNA(morphology, cytology, CEA(ng/ml)) with CT/MRI in the diagnosis of pancreatic cystic lesions. Surgical pathology is used as gold standard Established CEA cut-offs of >192 ng/ml were used for mucinous assessment and >1000 ng/ml for established cancer assessment. A CEA value of 5 ng/ml or less was indicative of a serous cyst

SECONDARY OUTCOMES:
Accuracy of EUS-FNA vs morphology | 10 years
  To compare the accuracy of EUS-FNA(morphology, cytology, CEA(ng/ml)) with EUS morphology alone in the diagnosis of pancreatic cystic lesions. Surgical pathology is used as gold standard.Established CEA cut-offs of >192 ng/ml were used for mucinous assessment and >1000 ng/ml for established cancer assessment. A CEA value of 5 ng/ml or less was indicative of a serous cyst
Accuracy of EUS FNA vs cytology | 10 years
  To compare the accuracy of EUS-FNA(morphology, cytology, CEA (ng/ml)) with EUS cytology alone in the diagnosis of pancreatic cystic lesions. Surgical pathology is used as gold standard.Established CEA cut-offs of >192 ng/ml were used for mucinous assessment and >1000 ng/ml for established cancer assessment. A CEA value of 5 ng/ml or less was indicative of a serous cyst
Accuracy of EUS FNA vs CEA | 10 years
  To compare the accuracy of EUS-FNA(morphology, cytology, CEA (ng/ml)) with EUS CEA(ng/ml) alone in the diagnosis of pancreatic cystic lesions. Surgical pathology is used as gold standard.Established CEA cut-offs of >192 ng/ml were used for mucinous assessment and >1000 ng/ml for established cancer assessment. A CEA value of 5 ng/ml or less was indicative of a serous cyst